CLINICAL TRIAL: NCT01221896
Title: Input of C11-Choline PET/CT in Localization of Parathyroid Adenoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: choline2010-HMO-CTIL
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Hyperparathyroidism
Keywords: Localization of a parathyroid adenoma in patients with primary hyperparathyroidism.
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hyperparathyroidism: Patients with hyperparathyroidism, prior to surgery.
  Interventions: Procedure: C11-Choline PET/CT

INTERVENTIONS:
Procedure: C11-Choline PET/CT

SUMMARY:
The purpose of the study is to determine a possible input of C11-Choline PET/CT in identification and localization of a parathyroid adenoma (PTA).

Preoperative localization of a PTA has been previously documented in multiple series, and is usually based on scintigraphy and on US.

Currently, the conventional technique for localization of a PTA is a dual-isotope scan with Tc99m-MIBI and Tc99m pertechnetate. This study is acquired over at least 3 hours, includes two i.v. injections and the patient has to stay 15-30 min per acquisition under the camera.

In addition, there is no anatomical imaging and further correlation with US is usually recommended.

In contrast, PET/CT study with C11-Choline takes as long as 10 min., includes one injection, and provides data of higher resolution of functional (PET) and anatomical imaging (CT).

Furthermore, dosimetric data shows that the total effective dose from Tc99mMIBI and Tc99m pertechnetate injection is (without CT): 0.5957 rem; and from C11-Choline injection and CT of a chest is: 0.3128 - 0.8628rem.

ELIGIBILITY:
Inclusion Criteria:

* Elevation of a calcium and parathyroid hormone in the serum

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with elevated PTH in search of a PTA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Improved localization of a parathyroid adenoma

SECONDARY OUTCOMES:
Facilitation of detection of the parathyroid adenoma at surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel